CLINICAL TRIAL: NCT05856188
Title: Efficacy of Glutamine in Management of Radiation Induced Mucositis in Patients With Head and Neck Cancer (A Randomized Controlled Clinical Study)
Brief Title: Efficacy of Glutamine in Management of Radiation Mucositis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Oral Mucositis
Record Dates: First submitted 2023-03-25; First posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Radiation-Induced Mucositis
Keywords: glutamine, Oral Mucositis, Salivary TGF b1
MeSH Terms: conditions — Stomatitis | interventions — Glutamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group I (Test group): (Experimental): Will include twenty patients receiving Glutamine oral suspension (5 grams of glutamine and 5 g maltodextrin dissolved in cold water) 30 min before a meal, 3 times per day through swish and swallow technique25 throughout the radiotherapy period.
  Interventions: Dietary Supplement: Glutamine
- Group II (Control group) (Placebo Comparator): Included twenty patients receiving maltodextrin oral suspension (5 g maltodextrin dissolved in cold water) 30 min before a meal, 3 times per day through swish and swallow technique throughout the radiotherapy period along with general measures as well as analgesic drugs according to the WHO scale.
  Interventions: Dietary Supplement: Glutamine

INTERVENTIONS:
Dietary Supplement: Glutamine — Biologic

SUMMARY:
The goal of this [ type of study: Clinical trial] is to test effectiveness of glutamine in management of Radiation Induced Mucositis in head and neck cancer patients.

The main question [s] ] is to [ learn about, test, compare etc.] it aims to answer are:

1. Is glutamine effective in management of Radiation Induced Mucositis?
2. Does Glutamine oral suspension affect the level of TGFβ1 in saliva of patients with radiation induced mucositis? participants will be asked to dissolve oral glutamine and maltodextrin in distalled water and swish and swallow three times daily during radiotherapy.

DETAILED DESCRIPTION:
Oral Mucositis (OM) refers to inflammation and ulceration of the oral mucosa as a side-effect of cancer therapy. OM and esophagitis can occur secondary to systemic chemotherapy for cancer, high-dose chemotherapy as a hematopoietic transplant preparative regimen or due to radiation therapy (RT) for head and neck (H&N) cancer or if the oropharynx or esophagus is in field during and after radiation of bone metastases. OM is a common problem and occurs in about 20-40% of patients receiving conventional chemotherapy for solid tumors, about 80% of patients receiving high dose chemotherapy prior to a hematopoietic stem cell transplantation (HSCT) and almost all patients receiving RT for H&N cancer. Ulcerative OM and esophagitis are extremely painful, with many patients needing systemic opioids such as morphine or fentanyl for pain management.1 Oral mucositis is an acute mucosal inflammation that starts as redness and progresses to an increased ulceration and pseudomembrane formation, which represent a temporary barrier until cellular repair promotes healing. The impaired mucosal tissue often permits bacteria and fungi to penetrate into damaged mucosa and cause infections.2 Mucositis is divided into 4 phases: an initial inflammatory/ vascular phase, an epithelial phase, an ulcerative/bacteriological phase, and a wound healing phase.3 In the initial stage, irradiation or chemotherapy, by producing free radicals and Reactive oxygen species (ROS), harmfully influences cells and strands of DNA in the basal epithelium and the submucosa and leads to lesions. ROS also activate transcription factors and leads to cell destruction in later stages. In the next stage, not only ROS but also damaged cells and DNA start a cascade of reactions. During these reactions, proinflammatory cytokines produce and lead to lesions and basal cell apoptosis. These products have a positive reaction as well, and strengthen the lesions. In this stage, the tissue appears to be normal, with only with slight erythema. In the third stage, painful lesions appear and are colonized by bacteria. Bacterial colonization can lead to the release of new pro-inflammatory cytokines. After stopping cancer treatment, oral mucositis vanishes little by little. In the healing process, symptoms decrease and the mucosa become normal, but outstanding neovascularization remains. This tissue is easily broken and it is susceptible to chemotherapy and/or radiotherapy in future periods of cancer treatments.4

. This diversity in scoring systems for Oral Mucositis may lead to controversies among studies. The most widely used measurements for oral mucositis are the World Health Organization(WHO) and Radiation Therapy Oncology Group (RTOG) scales as below.

Also, the Oral Mucositis Assessment Scale, and a Visual Analog Pain Scale (patient reporting scale of 0-10) are used for grading of mucositis. Mucosal changes like redness, ulceration with functional outcomes such as inability to eat and pain have been assessed in these scales. Based on clinical examination, 4 distinct grades can be determined for mucositis from 0 to 4 scores. Higher grades of mucositis (grade 3-4) are associated with loss of taste, hemorrhage, decreased intake of food and fluids, ulceration, pain, loss of voice, and low quality of life.5 The biomarkers can be considered promising tools for prediction and evaluation of oral mucositis. Eight groups of biomarkers were analyzed: growth factors, cytokines, acute-phase inflammatory markers, genetic factors, general proteins, plasma antioxidants and apoptotic proteins.6 Growth factors are proteins released by individual cells to transmit messages to other cells and to stimulate cellular growth, proliferation, and differentiation.7 Regarding the epithelia growth factor (EGF), it was observed a decrease in EGF levels during RT and a trend to reduced EGF in patients with more severe OM.8 Another important growth factor analyzed was the transforming growth factorβ (TGFβ), which controls cellular homeostasis and proliferation, wound healing, immunosuppression, and angiogenesis.9 It was observed that a TGFβ1 level was significantly higher in patients experiencing severe radiation toxicity, confirming that damaged tissues contribute to higher plasma TGFβ1 level.10 Cytokines are also involved in RT-induced mucositis because they are released by disintegrating cells or by an immune reaction, resulting in the recruitment of inflammatory cells and in the development of toxicity.11 It was observed that the level of interleukins IL-6, IL-10 and IL-1 β seemed to be related to severe mucositis.12 Acute-phase inflammatory markers are also used as biomarkers to predict the risk for patients developing OM as a consequence of cancer treatment. C-reactive protein (CRP) is one of these markers, and it contributes to body defense by neutralizing inflammatory agents and it can be easily measured as a quantitative marker of inflammatory activity.13 It was demonstrated an increase of CRP and correlation between this increase and the progression of mucositis. It could only observe during the initial weeks of treatment.11 Erythrocyte Sedimentation Rate (ESR) is another important marker of the acute-phase inflammatory response, used to evaluate benign inflammatory conditions and neoplastic diseases. An increase in ESR levels during cancer treatment was observed, followed by a decrease in concentration of this biomarker. This variation was related to the grading of mucositis, which also initially increased in severity and then decreased towards the end of treatment.14 Glutamine is an L-alpha-amino acid. It is the most abundant free amino acid in human blood. Glutamine is needed for several functions in the body including for the synthesis of proteins as well as an energy source. Glutamine can be synthesized by the body and can also be obtained from the diet if needed.15 Glutamine is an important nitrogen donor in intracellular metabolism and in the maintenance of intestinal tract, immune cells, and muscle.16 Weight loss in cancer patients is common, but sarcopenia (loss of muscle mass) is associated with increased complications and significantly worse survival.17 Glutamine is a preferred fuel for both lymphocytes and gastrointestinal (GI) tract 18, thus it plays an important role in helping to defend against infections and to assist mucosa in being a barrier against infection.

Glutamine has a central role in intracellular metabolism and acts as a nitrogen shuttle between muscle and other tissues; it is at a high and relatively stable concentration in plasma and red blood cells and at a much higher concentration in muscle compared to other amino acids.19 Since plasma glutamine concentrations are only minimally affected over time by either glutamine ingestion or infusion, muscle can be considered as a "bank" and the liver can be considered as the "banker".17 Neutrophils, macrophages, and lymphocytes are needed for mucosal barrier immune defenses. Since glutamine is fuel for leukocytes, topical/oral/enteral glutamine may contribute to mucosal healing by not only a direct effect on mucosal epithelial cells, but also by improvement in host mucosal immune function and ability to resist microbial invasion.16 Interestingly, resilience of lymphocyte recovery, as measured by absolute lymphocyte count (ALC) after the very first cycle of chemotherapy, has been associated with a better prognosis in a variety of malignancies including acute lymphoblastic leukemia as well as tumors such as osteosarcoma, Ewing sarcoma, and rhabdomyosarcoma . It is possible that better nutrition, with amino acids including glutamine as fuel for lymphocytes, could contribute to ALC recovery and/or resilience. Animal models and human studies have shown glutamine supplementation improves the ability to resist the toxic effects of radiation to the GI tract.15 Detoxification and resilience to free radical damage by chemotherapy (e.g., doxorubicin or cyclophosphamide) and/or radiation of normal tissues and tumors can involve the antioxidant glutathione. Since glutamine is a substrate for glutathione synthesis, adequate mucosal cell glutamine may contribute towards improved healing after chemotherapy and radiation damage 20 as well as, interestingly, the simultaneous inhibition of glutathione levels in tumors, too.21 Furthermore, decreased inflammatory cytokines in normal cells and increased pro-apoptosis proteins in cancer cells were observed with glutamine + disaccharide supplementation. Thus, glutamine can contribute to selective improvement in host cell resilience, less inflammation, and decreased ability of tumors to detoxify chemotherapy or resist radiation, i.e. an improved therapeutic index of the anti-cancer therapy.22 Glutamine can be administrated by three common routes; parental, oral and topical through swishing. Topical oral swish and swallow glutamine has potential to ameliorate not only OM, but also esophagitis and enteritis after cancer chemotherapy and radiation. A small amino acid intervention may make a difference and possibly contribute to better overall nutritional status, improved survival with fewer complications, and ultimately less sarcopenia and lymphopenia.15 To the moment , there are no published studies regarding assessment of salivary TGFβ1 in glutamine treatment of radiotherapy induced mucositis So regarding the forementioned properties of glutamine, The hypothesis is to assess if the glutamine could affect severity of mucositis and the level of salivary TGFβ1.

The purpose of this study is to evaluate the influence of glutamine in treatment of radiation induced mucositis in head and neck cancer patients and measuring the TGFβ salivary level before and after treatment with glutamine.

ELIGIBILITY:
Inclusion Criteria:

* a) Patients with a confirmed histologic diagnosis of H&N malignancy who are referred to non-palliative radiotherapy in the oral cavity.

  b) Patient who is receiving radiation therapy with intensity modified radiotherapy IMRT or 3D techniques.

  c) Patients received 50-70 Gy of total radiation at the rate of 2 Gy/fraction daily and 5 fractions/week.

  d) Patient who received concurrent chemotherapy with radiotherapy e) Presence of Oral Mucositis f) Age 20-70 years old g) Willing to participate in the study h) Able to complete the study assessments

Exclusion Criteria:

* a) Have a confirmed or medically treated diabetes mellitus25 b) Radiotherapy within the last 6 months prior to this study c) Vulnerable patients

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Change from World Health Organization Oral Toxicity Scale Grading of Oral Mucositis during radiotherapy. | Two points: -"baseline which is at the second week of radiotherapy" while -"the end of the radiotherapy is at seventh week of the radiotherapy or 4-5 weeks from baseline.
  World Health Organization Oral Toxicity Scale Grading of Oral Mucositis ranges from "1,2,3,4) the grade1 means the least clinical sign and symptoms while grade 4 means the worst clinical sign and symptoms of mucositis.
Change in the level of salivary transforming growth factor beta 1 during radiotherapy. | Two points: -"baseline which is at the second week of radiotherapy" while -"the end of the radiotherapy is at seventh week of the radiotherapy or 4-5 weeks from baseline.
  salivary level of transforming growth factor beta 1 assessment using enzyme linked immune assay may range from 10-4000ng/L

SECONDARY OUTCOMES:
Change in Pain visual analog scale during radiotherapy. | Two points: -"baseline which is at the second week of radiotherapy" while -"the end of the radiotherapy is at seventh week of the radiotherapy or 4-5 weeks from baseline.
  Pain visual analog scale range from (0 to 10
  ), 0 means no pain felt, while 10 means the worst unbearable pain.

CONTACTS AND LOCATIONS:
Overall Officials: Suzan SA Ibrahim, professor, Study Director — faculty of Dentistry- Ainshams university
Locations (2):
- Egypt (2):
  - ain shams University, Cairo
  - Fatma E.Sayed, Cairo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Arutla M, Raghunath M, Deepika G, Jakkampudi A, Murthy HVV, Rao GV, Reddy DN, Talukdar R. Efficacy of enteral glutamine supplementation in patients with severe and predicted severe acute pancreatitis- A randomized controlled trial. Indian J Gastroenterol. 2019 Aug;38(4):338-347. doi: 10.1007/s12664-019-00962-7. Epub 2019 Oct 14. PMID 31612309
- [Result] Fahr MJ, Kornbluth J, Blossom S, Schaeffer R, Klimberg VS. Harry M. Vars Research Award. Glutamine enhances immunoregulation of tumor growth. JPEN J Parenter Enteral Nutr. 1994 Nov-Dec;18(6):471-6. doi: 10.1177/0148607194018006471. PMID 7602720
- [Derived] Ibrahim SS, Hassanein FEA, Zaky HW, Gamal H. Clinical and biochemical assessment of the effect of glutamine in management of radiation induced oral mucositis in patients with head and neck cancer: Randomized controlled clinical trial. J Stomatol Oral Maxillofac Surg. 2024 Jun;125(3S):101827. doi: 10.1016/j.jormas.2024.101827. Epub 2024 Mar 15. PMID 38493953